CLINICAL TRIAL: NCT06845007
Title: PROMBot: a Web Platform for Collecting Patient-Reported Outcome Measures Via a Chatbot
Brief Title: PROMBot: a Web Platform for Collecting Outcomes for Hypertension Patients Via a Chatbot
Status: Recruiting | Type: Observational
Sponsor: Ana Rita Londral (Other)
Responsible Party: Sponsor-Investigator, Ana Rita Londral, Investigator, Value for Health CoLAB
Organization: Value for Health CoLAB (Other)
Other Study IDs: VOH_PROMBOT
Record Dates: First submitted 2025-02-06; First posted 2025-02-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: Chatbot; Web plataform; PROMBot; Patient Monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hypertension Group: This study includes only one group. This group will consist of patients with hypertension, and after a patient is identified, they will be followed up using the PROMBot platform for the subsequent 12 weeks. In the first week, the patient will be required to record their diastolic and systolic blood pressure values daily and answer a quiz on hypertension-related topics. In the second week, the participant will continue recording their blood pressure values, but only every other day. From the third to the tenth week, the participant may choose to receive tips on nutrition recipes and exercises they can perform to increase physical activity. In the 11th week, the participant will again measure their blood pressure, but the values will only be recorded on the 1st, 3rd, 5th, and 7th days. Finally, in the 12th week, the participant will resume recording daily blood pressure values in PROMBot.

SUMMARY:
The present study is observational and aims to evaluate the PROMBot service in managing patients' hypertension, simplify the follow-up process, and empower patients to actively participate in their own care.

DETAILED DESCRIPTION:
In the last two decades, research and development (R&D) efforts in remote patient monitoring (RPM) technologies have primarily focused on the technical challenges of providing care in unconventional settings. Several pilot initiatives have emerged, ranging from chronic disease management to episodic care, such as post-surgical follow-ups, to leverage the advantages of RPM. These benefits include improving the continuity of outpatient care, enabling more informed health decision-making, anticipating complications, and reducing costs. For instance, in the context of post-surgical follow-up, RPM has demonstrated significant potential in reducing severe complications and increasing patient safety during the critical period following hospital discharge. By enabling healthcare professionals to continuously monitor clinical indicators and patient-reported outcome measures (PROMs), RPM plays a vital role in ensuring effective surveillance.

A systematic review highlights evidence that chatbots could be effective tools for increasing physical activity, fruit and vegetable consumption, and improving sleep duration and quality. In a recent study, users of a chatbot for hypertensive patients demonstrated greater knowledge and skills in blood pressure (BP) monitoring and slightly better accuracy in BP measurements.

However, there is still little research on implementation studies. After the COVID-19 pandemic, there was an increase in demand for RPM-based services due to postponed surgeries and the shift from in-person to remote care. As a result, ongoing pilot initiatives increased without sufficient planning. This lack of time and resources poses risks to both accessibility and care quality. Research is needed to explore the characteristics of different RPM systems that drive high-value RPM services.

Existing literature consistently emphasizes three key components for an effective RPM system: care team organization, technology utilization, and patient engagement activities. Therefore, using participatory action research (PAR) methodologies, where clinical teams and patients are actively involved in the research, becomes essential to ensure that the technological solutions developed and deployed align with the needs and preferences of end users, thereby maximizing solution adoption.

The PROMBot was created using a PAR approach, incorporating feedback from various stakeholders, including patients, healthcare professionals, software developers, and researchers. This collaborative effort allowed for the suggestion, testing, and evaluation of the platform's functionalities, ensuring both effectiveness and usability. By adopting a PAR approach, the development and implementation of the PROMBot platform addressed real-world challenges and requirements associated with implementing digital health services.

This study will last for 6 months and aims to evaluate the PROMBot service The implementation of the PROMBot platform in CUF's services serves two primary purposes: 1) to help CUF design and assess various remote follow-up interventions, and 2) to explore different use cases for the application of PROMBot By leveraging PROMBot, patients will have the ability to conveniently record their health parameters and symptoms daily Additionally, the platform will provide a user-friendly digital interface that supports care teams throughout the follow-up process.

This study is an observational study that will contribute to the exploration of different use cases for the implementation of innovative patient-centered systems, potentially positioning the patient monitoring service as a model to be followed by other clinical departments, both nationally and internationally By using technology and remote monitoring, this study aims to enhance patient care and set new standards for remote follow-up in the context of CUF, improving outcomes and promoting patient-centered healthcare practices.

The specific objectives of this study are:

1. To obtain a more continuous blood pressure history to personalize healthcare
2. To provide information to healthcare professionals about the knowledge acquired by the patient regarding the behavior to adopt
3. To evaluate improvements in participants' health-related knowledge and behaviors, such as salt consumption, physical exercise practices, medication adherence, and preparation of healthy meals
4. To study patient engagement levels with the chatbot and assess treatment adherence throughout the program
5. To evaluate the ease of use and perception of usefulness of the chatbot by participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old.
* Diagnosed with hypertension, based on ICD-9 codes (401-401.9).
* Independent in performing activities of daily living.
* Ability to respond to SMS messages.

Exclusion Criteria:

* Diagnosis of Parkinson's disease.
* Refusal to sign the informed consent form.
* Diagnosis of cancer.
* Mobility limitations that prevent engaging in physical activity.
* Lack of a smartphone with internet access.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants must have hypertension, live in Portugal and be followed by a doctor at the CUF hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview | After interacting with the chatboot, which took place over 12 weeks.
  The semi-structured interviews will be conducted by the research team and aim to gather participants' reactions and experiences with the chatbot. The questions included in the interview are:
  1. Do you consider PROMBot easy to use?
  2. Do you consider PROMBot useful? Please answer yes or no.
  3. Which types of messages from PROMBot were the most useful for you?
  4. What improvements would you suggest for PROMBot?
  5. Was interacting with PROMBot enjoyable?
  6. Would you like to continue using PROMBot to record your blood pressure values? Why? Please briefly justify your reasons for wanting to continue or not.
  7. Would you like to continue using PROMBot to receive medication reminders? Why? Please briefly justify your reasons for wanting to continue or not.
  8. Would you like to continue using PROMBot to receive tips on healthy habits? Why? Please briefly justify your reasons for wanting to continue or not.

SECONDARY OUTCOMES:
Engagement | After interacting with the chatboot, which took place over 12 weeks.
  The level of patient engagement will be measured by calculating a proxy based on the number of messages sent to the chatbot.
Treatment Adherence | After interacting with the chatboot, which took place over 12 weeks.
  The level of treatment adherence will be measured by calculating a proxy based on the number of messages sent following blood pressure measurements by the patient.
Health Literacy | After interacting with the chatboot, which took place over 12 weeks.
  During the program, patients will be assessed on their knowledge of health literacy content related to hypertension in the following areas (self-reported):
  Health Literacy Knowledge Assessment on Hypertension Topics:
  Salt Consumption; Engagement in Physical Exercise.
  The questions will be multiple choice, with one correct answer for each question.
Intra-Individual Effects | After interacting with the chatboot, which took place over 12 weeks.
  To evaluate the intra-individual effect of using PROMBot, participants will be invited to respond to four questions before and one week after the program to assess salt consumption habits, frequency of blood pressure measurement, and physical activity:
  Question 1:
  In the past week, how many days did you engage in physical exercise or any physical activity for 30 minutes or more?
  Possible response:
  0 - None, 1 - 1 day, 2 - 2 days, 3 - 3 days, 4 - 4 days, 5 - 5 days, 6 - 6 days, 7 - 7 days.
  Question 2:
  In the past week, how many days did you record your blood pressure?
  Possible response:
  0 - None, 1 - 1 day, 2 - 2 days, 3 - 3 days, 4 - 4 days, 5 - 5 days, 6 - 6 days, 7 - 7 days.
  The minimum value on this scale is 0 and the maximum value is 7. A higher score means a better result.
Intra-Individual Effects | After interacting with the chatboot, which took place over 12 weeks.
  To evaluate the intra-individual effect of using PROMBot, participants will be invited to respond to four questions before and one week after the program to assess salt consumption habits, frequency of blood pressure measurement, and physical activity:
  Question 3:
  In the past week, how often did you add salt to your food?
  Possible response (Likert scale):
  1 - Never or almost never, 2 - Sometimes, 3 - Most of the time, 4 - Always.
  The minimum value on this scale is 0 and the maximum value is 4. A higher score means a worse result.
Intra-Individual Effects | After interacting with the chatboot, which took place over 12 weeks.
  To evaluate the intra-individual effect of using PROMBot, participants will be invited to respond to four questions before and one week after the program to assess salt consumption habits, frequency of blood pressure measurement, and physical activity:
  Question 4:
  In the past week, how often did you take your blood pressure medication as prescribed by your doctor?
  Possible response:
  1 - Never, 2 - Rarely, 3 - Sometimes, 4 - Always.
  The minimum value on this scale is 0 and the maximum value is 4. A higher score means a better result.

OTHER OUTCOMES:
Gender | Before the interaction with the chatboot begins
  Personal Identification : Gender, Male / Female
Age | Before the interaction with the chatboot begins
  Personal Identification : Age (years).
Education Level | Before the interaction with the chatboot begins
  Personal Identification : Education Level.
Primary Diagnosis | Before the interaction with the chatboot begins
  Current Condition: Primary Diagnosis: Essential high blood pressure; Secondary high blood pressure
Blood Pressure | Before the interaction with the chatboot begins
  Current Condition: Blood Pressure (Systolic and diastolic) values recorded throughout the program.
Behavioral assessment - Medication | Before the interaction with the chatboot begins
  Number of days the patient adhered to prescribed medication during the program (number of days).
  Na primeira semanas perguntamos 2 vezes ao dia (dia e noite). Na 2ª senana, 1º 4º 7º. nas semanas de intervalo pode receber ou não
Physical exercise engagement | Before the interaction with the chatboot begins
  Days on which the patient requested information about exercise (number of days)
Healthy recipes engagement | Before the interaction with the chatboot begins
  Days on which the patient requested information about exercise (number of days)

CONTACTS AND LOCATIONS:
Locations (1):
- CUF, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farias FAC, Dagostini CM, Bicca YA, Falavigna VF, Falavigna A. Remote Patient Monitoring: A Systematic Review. Telemed J E Health. 2020 May;26(5):576-583. doi: 10.1089/tmj.2019.0066. Epub 2019 Jul 17. PMID 31314689
- [Background] Echeazarra L, Pereira J, Saracho R. TensioBot: a Chatbot Assistant for Self-Managed in-House Blood Pressure Checking. J Med Syst. 2021 Mar 15;45(4):54. doi: 10.1007/s10916-021-01730-x. PMID 33723721
- [Background] Singh B, Olds T, Brinsley J, Dumuid D, Virgara R, Matricciani L, Watson A, Szeto K, Eglitis E, Miatke A, Simpson CEM, Vandelanotte C, Maher C. Systematic review and meta-analysis of the effectiveness of chatbots on lifestyle behaviours. NPJ Digit Med. 2023 Jun 23;6(1):118. doi: 10.1038/s41746-023-00856-1. PMID 37353578
- [Background] Park DK, Jung EY, Park RW, Lee YH, Hwang HJ, Son IA, Hu MH. Telecare system for cardiac surgery patients: implementation and effectiveness. Healthc Inform Res. 2011 Jun;17(2):93-100. doi: 10.4258/hir.2011.17.2.93. Epub 2011 Jun 30. PMID 21886870
- [Background] Pekmezaris R, Mitzner I, Pecinka KR, Nouryan CN, Lesser ML, Siegel M, Swiderski JW, Moise G, Younker R Sr, Smolich K. The impact of remote patient monitoring (telehealth) upon Medicare beneficiaries with heart failure. Telemed J E Health. 2012 Mar;18(2):101-8. doi: 10.1089/tmj.2011.0095. Epub 2012 Jan 27. PMID 22283360
- [Background] Baginski BN, Byrne KA, Vaz DG, Barber R, Blackhurst D, Tibbett TP, Guichard JL. Development and implementation of a remote patient monitoring program for heart failure: a single-centre experience. ESC Heart Fail. 2021 Apr;8(2):1349-1358. doi: 10.1002/ehf2.13214. Epub 2021 Jan 27. PMID 33503681
- [Background] Pare G, Jaana M, Sicotte C. Systematic review of home telemonitoring for chronic diseases: the evidence base. J Am Med Inform Assoc. 2007 May-Jun;14(3):269-77. doi: 10.1197/jamia.M2270. Epub 2007 Feb 28. PMID 17329725
- [Background] Vegesna A, Tran M, Angelaccio M, Arcona S. Remote Patient Monitoring via Non-Invasive Digital Technologies: A Systematic Review. Telemed J E Health. 2017 Jan;23(1):3-17. doi: 10.1089/tmj.2016.0051. Epub 2016 Apr 26. PMID 27116181